CLINICAL TRIAL: NCT06322433
Title: Long Term Follow-up of Eyes With High Myopia
Brief Title: Follow up of High Myopic Eyes
Acronym: FWUPMIOPIA_ E
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 37C301
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pathologic Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: no drugs used for this study — tomographic, angiographic and clinical follow up

SUMMARY:
In this non-interventional retrospective and prospective observational study, the long-term evolution of clinical and iconographic characteristics of patients with pathological myopia will be considered Changes of some specific clinical, tomographic and angiographic variables evaluated on the baseline and after a minimum of 5 years follow-up will be studied.

ELIGIBILITY:
Inclusion Criteria:

- high myopia

Exclusion Criteria:

* acute ischemic optic neuropathy
* macular and peripapillary atrophy
* other forms of maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of patients presenting at our Institution with eye myopia
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with neovascularization at follow-up visit | at 5 years of follow up
  Evaluation of choroidal neovascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy